CLINICAL TRIAL: NCT03442192
Title: A Comparative Effectiveness Demonstration Project for Linkage and Retention in PrEP Care for Men Who Have Sex With Men (PCA)
Brief Title: A Comparative Effectiveness Demonstration Project for Linkage and Retention in PrEP Care for Men Who Have Sex With Men
Acronym: PCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID erupted and change in policy making all visits throughout hospital telemedicine
Sponsor: Johns Hopkins University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00132612
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Adherence, Patient
Keywords: PrEP; virtual; adherence; retention
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Changed from randomization to provide PrEP Care Anywhere approach to everyone enrolled to determine differences in engagement, retention and adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP Care Anywhere Services (Other): The PrEP Care Anywhere intervention adapts peer PrEP case management for virtual delivery and provides clinical services through a tele-health program, delivered by the same clinic providers. After an initial face-to-face intake clinical evaluation within the clinic, will then receive the remaining PrEP clinical evaluations via telemedicine using the HIPPA compliant polycom platform. Case management interventions will be conducted virtually via the PrEPme application, telephone consultation, text, or email.
  Interventions: Other: PrEP Care Anywhere Services

INTERVENTIONS:
Other: PrEP Care Anywhere Services — PrEP Virtual Clinic Visits. PrEP clinical care will follow guidelines as established by the CDC for PrEP clinical evaluation and follow-up. Appointments will be set up in the same process as any practice visit and require the same clinical documentation and billing requirements, but will have a separate clinic designation for the visit type. At any time during the study, a patient can request a face-to-face visit with the provider. The provider may also request a face-to-face visit based on patient presentation and/or laboratory results.
  The typical visit options will include:
  * On demand peer interim visits- participants can text, chat (via PrEPme app) or call to access an on demand virtual support visit with a peer Case Manager (CM).
  * HIV and Sexually Transmitted Infection (STI) at Home Self-Testing

SUMMARY:
This research is being done to learn more about the differences in engaging, recruiting, linking and adhering to pre-exposure prophylaxis (PrEP) services for men who have sex with other men at risk for HIV in Baltimore City.

In 2012, the U.S. Food and Drug Administration (FDA) approved the use of Truvada as pre-exposure prophylaxis (PrEP) to help prevent HIV infection. In the intervention, a virtual, PrEP Care Anywhere Telemedicine approach supported by virtual peer-navigator will be compared to standard clinic-based PrEP services with face-to-face peer navigation. The study will evaluate whether PrEP Care Anywhere, which is more patient-centered, will improve adherence and retention in PrEP care.

DETAILED DESCRIPTION:
According to the Centers for Disease Control and Prevention (CDC), the estimated lifetime risk for HIV is 1 in 2 for Black men who have sex with men (MSM) and 1 in 4 for Latino MSM. In 2012, the U.S. Food and Drug Administration approved the use of Truvada as pre-exposure prophylaxis (PrEP) to help prevent HIV infection. However, PrEP uptake and adherence among MSM of color in particular remains low. Part of the challenge of increasing PrEP uptake and adherence among MSM of color is related to a historical lack of ethnic and sexual minority engagement in health care systems, perceptions of racism and negativity, and inequities in treatment.

In order to engage, recruit, link, and retain MSM at substantial risk of HIV infection, this study proposes a randomized controlled pilot trial among 100 HIV-negative MSM of color (50 per arm) in Baltimore City to determine differences in engagement, retention and adherence to Truvada along with PrEP services. In the intervention, a virtual, PrEP Care Anywhere Telemedicine approach supported by virtual peer-navigator will be compared to standard clinic-based PrEP services with face-to-face peer navigation. The study will evaluate whether PrEP Care Anywhere, as a more client-centered approach, will improve adherence and retention.

The specific aims of the Randomized Controlled Trial (RCT) pilot are:

* To explore differences in linkage, engagement (uptake) and retention in PrEP services between traditional clinic-based PrEP services compared to the PrEP Care Anywhere (i.e., virtual) approach

Secondary Objectives

* To describe engagement with the smartphone application, PrEP me, in the PrEP Care Anywhere arm
* To evaluate the feasibility and scalability of the intervention package by measuring the number of peer intervention contacts (e.g., text message, email, phone, in person, mobile app chats) per participant over 12 months
* To evaluate biological markers of adherence among a subset of HIV-negative participants and all participants who seroconvert
* To evaluate agreement in self-reported daily adherence (app-based reporting) to standard quarterly clinic-based self-report and to correlate self-reported adherence with biomarkers of adherence including peripheral blood mononuclear cells (PBMC) and plasma levels of tenofovir disoproxil fumarate (TDF) in a subset of participants
* To compare longitudinal changes in sexual risk behavior, health care utilization, intimate partner violence, stigma, substance use and mental health between the two study arms over 12 months by administering questionnaires at baseline, month 1 and quarterly visits
* To assess feasibility and acceptability of virtual self-testing for HIV and sexually transmitted infections
* To compare the experience of and satisfaction with linkage to and engagement in ongoing HIV prevention services among participants by conducting and analyzing exit interviews

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older who are HIV-negative and meeting CDC risk criteria
* Persons self-identifying as Black/African American, Latino or other men of color up to 20% Caucasian
* Men who report unprotected sex with another male partner in preceding twelve months
* Expressed interest in seeking HIV PrEP clinical services
* Willing to participate in study-related procedures, including baseline and study visits every three months
* Willing and able (i.e., access to internet connectivity) to participate in virtual PrEP model through EPIC, polycom platform
* Insured with plan that is accepted by Johns Hopkins (study team will conduct monthly tracking of insurance plans accepted by the Bartlett Specialty Care Clinic)
* Willing to receive PrEP care at Johns Hopkins

Exclusion Criteria:

* Under 18 years of age
* Unable to read, write or speak English
* For medical reasons, are unable to receive TDF/FTC for PrEP (including HIV- positive persons)
* Participating in another PrEP clinical trial or HIV vaccination study
* Not insured with a plan that is accepted at Johns Hopkins
* Not willing or able (i.e. access to internet connectivity) to participate in virtual PrEP model
* Not willing to receive PrEP care at Johns Hopkins

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — men who have sex with men (MSM)
Enrollment: 20 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
PrEP Uptake | 1 month
  Primary outcome 1 will examine PrEP uptake at Month 1, among those not already taking PrEP at baseline, defined as Tenofovir (TFV) levels of 35.5 ng/mL or greater, using students T-test

SECONDARY OUTCOMES:
PrEP Adherence | 12 months
  Adherence at Month 12, defined as persistent TFV levels of 35.5 ng/mL between the arms will be evaluated by Cox Proportional Hazard models

OTHER OUTCOMES:
PrEP Retention | Month 3, 6 and 9 months
  Retention will be tested at 3, 6 and 9 months using chi-square test to compare retention between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Farley, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirby T, Thornber-Dunwell M. Uptake of PrEP for HIV slow among MSM. Lancet. 2014 Feb 1;383(9915):399-400. doi: 10.1016/s0140-6736(14)60137-9. No abstract available. PMID 24494225
- [Background] Arnold EA, Rebchook GM, Kegeles SM. 'Triply cursed': racism, homophobia and HIV-related stigma are barriers to regular HIV testing, treatment adherence and disclosure among young Black gay men. Cult Health Sex. 2014 Jun;16(6):710-22. doi: 10.1080/13691058.2014.905706. Epub 2014 May 2. PMID 24784224
- [Background] Cahill S, Taylor SW, Elsesser SA, Mena L, Hickson D, Mayer KH. Stigma, medical mistrust, and perceived racism may affect PrEP awareness and uptake in black compared to white gay and bisexual men in Jackson, Mississippi and Boston, Massachusetts. AIDS Care. 2017 Nov;29(11):1351-1358. doi: 10.1080/09540121.2017.1300633. Epub 2017 Mar 12. PMID 28286983
- [Background] Freeman R, Gwadz MV, Silverman E, Kutnick A, Leonard NR, Ritchie AS, Reed J, Martinez BY. Critical race theory as a tool for understanding poor engagement along the HIV care continuum among African American/Black and Hispanic persons living with HIV in the United States: a qualitative exploration. Int J Equity Health. 2017 Mar 24;16(1):54. doi: 10.1186/s12939-017-0549-3. PMID 28340589
- [Background] Beck C, McSweeney JC, Richards KC, Roberson PK, Tsai PF, Souder E. Challenges in tailored intervention research. Nurs Outlook. 2010 Mar-Apr;58(2):104-10. doi: 10.1016/j.outlook.2009.10.004. PMID 20362779
- [Background] Hendrix CW, Chen BA, Guddera V, Hoesley C, Justman J, Nakabiito C, Salata R, Soto-Torres L, Patterson K, Minnis AM, Gandham S, Gomez K, Richardson BA, Bumpus NN. MTN-001: randomized pharmacokinetic cross-over study comparing tenofovir vaginal gel and oral tablets in vaginal tissue and other compartments. PLoS One. 2013;8(1):e55013. doi: 10.1371/journal.pone.0055013. Epub 2013 Jan 30. PMID 23383037
- [Background] DiFrancesco R, Rosenkranz SL, Taylor CR, Pande PG, Siminski SM, Jenny RW, Morse GD. Clinical pharmacology quality assurance program: models for longitudinal analysis of antiretroviral proficiency testing for international laboratories. Ther Drug Monit. 2013 Oct;35(5):631-42. doi: 10.1097/FTD.0b013e31828f5088. PMID 24052065
- [Background] Hendrix CW, Andrade A, Bumpus NN, Kashuba AD, Marzinke MA, Moore A, Anderson PL, Bushman LR, Fuchs EJ, Wiggins I, Radebaugh C, Prince HA, Bakshi RP, Wang R, Richardson P, Shieh E, McKinstry L, Li X, Donnell D, Elharrar V, Mayer KH, Patterson KB. Dose Frequency Ranging Pharmacokinetic Study of Tenofovir-Emtricitabine After Directly Observed Dosing in Healthy Volunteers to Establish Adherence Benchmarks (HPTN 066). AIDS Res Hum Retroviruses. 2016 Jan;32(1):32-43. doi: 10.1089/AID.2015.0182. Epub 2015 Oct 15. PMID 26414912
- [Background] Liu AY, Yang Q, Huang Y, Bacchetti P, Anderson PL, Jin C, Goggin K, Stojanovski K, Grant R, Buchbinder SP, Greenblatt RM, Gandhi M. Strong relationship between oral dose and tenofovir hair levels in a randomized trial: hair as a potential adherence measure for pre-exposure prophylaxis (PrEP). PLoS One. 2014 Jan 8;9(1):e83736. doi: 10.1371/journal.pone.0083736. eCollection 2014. PMID 24421901
- [Background] Castro FG, Barrera M Jr, Martinez CR Jr. The cultural adaptation of prevention interventions: resolving tensions between fidelity and fit. Prev Sci. 2004 Mar;5(1):41-5. doi: 10.1023/b:prev.0000013980.12412.cd. PMID 15058911
- [Background] Montgomery MC, Oldenburg CE, Nunn AS, Mena L, Anderson P, Liegler T, Mayer KH, Patel R, Almonte A, Chan PA. Adherence to Pre-Exposure Prophylaxis for HIV Prevention in a Clinical Setting. PLoS One. 2016 Jun 22;11(6):e0157742. doi: 10.1371/journal.pone.0157742. eCollection 2016. PMID 27333000
- [Background] Zheng JH, Rower C, McAllister K, Castillo-Mancilla J, Klein B, Meditz A, Guida LA, Kiser JJ, Bushman LR, Anderson PL. Application of an intracellular assay for determination of tenofovir-diphosphate and emtricitabine-triphosphate from erythrocytes using dried blood spots. J Pharm Biomed Anal. 2016 Apr 15;122:16-20. doi: 10.1016/j.jpba.2016.01.038. Epub 2016 Jan 21. PMID 26829517
- [Background] Whetten K, Reif S, Swartz M, Stevens R, Ostermann J, Hanisch L, Eron JJ Jr. A brief mental health and substance abuse screener for persons with HIV. AIDS Patient Care STDS. 2005 Feb;19(2):89-99. doi: 10.1089/apc.2005.19.89. PMID 15716640
- [Background] Wilson IB, Fowler FJ Jr, Cosenza CA, Michaud J, Bentkover J, Rana A, Kogelman L, Rogers WH. Cognitive and field testing of a new set of medication adherence self-report items for HIV care. AIDS Behav. 2014 Dec;18(12):2349-58. doi: 10.1007/s10461-013-0610-1. PMID 24077970